CLINICAL TRIAL: NCT07165028
Title: A Master Protocol for a Randomized, Controlled, Clinical Trial of Multiple Pharmacologic Agents in Adult Participants With Metabolic Dysfunction-Associated Steatotic Liver Disease Who Are at Increased Risk of Developing Major Adverse Liver Outcomes
Brief Title: A Master Protocol of Multiple Agents in Adults With Metabolic Dysfunction-Associated Steatotic Liver Disease (SYNERGY-Outcomes)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27610; 2025-522674-36-00 (EU CTIS Number); N1T-MC-MALO (Other: Eli Lilly and Company); N1T-MC-TZ01 (Other: Eli Lilly and Company); N1T-MC-RT01 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-08-28; First posted 2025-09-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Nonalcoholic Steatohepatitis; NASH; Fatty Liver; Fatty Liver Disease; SLD; Metabolic Dysfunction-Associated Fatty Liver Disease; MAFLD; Non-alcoholic Fatty Liver Disease; NAFLD; Hepatic Steatosis; Liver Related Outcomes; GLP1; Incretin; Non-Invasive Test
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Tirzepatide; retatrutide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tirzepatide (TZ01) (Experimental): Participants will receive tirzepatide subcutaneously (SC)
  Interventions: Drug: Tirzepatide
- Placebo (TZ01) (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo
- Retatrutide (RT01) (Experimental): Participants will receive retatrutide SC
  Interventions: Drug: Retatrutide
- Placebo (RT01) (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide (TZ01)
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide (RT01)
Drug: Placebo — Administered SC
  Arms: Placebo (RT01); Placebo (TZ01)

SUMMARY:
The main purpose of the SYNERGY-OUTCOMES study is to find out whether retatrutide and tirzepatide can prevent major adverse liver outcomes (MALO) in people with high-risk metabolic dysfunction-associated steatotic liver disease (MASLD). The study will enroll adults who have MASLD based on non-invasive tests (NITs), which indicate they are more likely to develop MALO. Participants will be randomly assigned within a Master Protocol to receive either retatrutide (N1T-MC-RT01), tirzepatide (N1T-MC-TZ01) or placebo. The trial plans to enroll about 4,500 adults and will run for approximately 224 weeks. Participants may have up to approximately 25 to 30 clinic visits throughout the study to monitor their health, complete study procedures, and assess liver function and disease progression.

Once the study is complete, eligible participants may participate in an optional 2-year extension study, in which all participants will receive either retatrutide or tirzepatide, even if they received placebo in the main study.

ELIGIBILITY:
Inclusion Criteria:

* Have liver fat content ≥8%
* Have ELF score of ≥9 and ≤10.8 at screening
* Have VCTE LSM ≥10 kilopascal (kPa) and <20 kPa at screening

Exclusion Criteria:

* Have any other type of liver disease other than MASLD
* Have a body mass index (BMI) <25 kilogram per square meter (kg/m2)
* Prior decompensated liver disease (history of esophageal/gastric varices, ascites, hepatic encephalopathy)
* Have lost more than 11 pounds within the 3 months prior to screening
* Have a hemoglobin A1c (HbA1c) greater than 10%
* Have type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Any Component of the Composite Endpoint for Major Adverse Liver Outcomes (MALO) | Baseline up to Study Completion (about 224 weeks)
  Composite endpoint comprised of progression to cirrhosis, development of large esophageal varices, gastric varices or development of varices needing treatment, development of ascites, development of hepatic encephalopathy, evidence of active or recent variceal hemorrhage, increase in model for end-stage liver disease (MELD) from ≤12 to ≥15, liver transplantation, all-cause mortality

SECONDARY OUTCOMES:
Change from Baseline in Enhanced Liver Fibrosis (ELF) Score | Baseline, Week 104
Change from Baseline in Vibration-Controlled Transient Elastography Liver Stiffness Measurement (VCTE LSM) | Baseline, Week 104
Percent Change from Baseline in Liver Fat Content (LFC) | Baseline, Week 104
Time to Occurrence of Progression to Cirrhosis | Baseline up to Study Completion (about 224 weeks)
Change from Baseline in Aspartate Aminotransferase (AST) | Baseline, Study Completion (about 224 weeks)
Change from Baseline in Alanine Aminotransferase (ALT) | Baseline, Study Completion (about 224 weeks)
Change from Baseline in Body Weight | Baseline, Study Completion (about 224 weeks)
Change from Baseline in Non-Alcoholic Steatohepatitis-CHECK Score (NASH-CHECK) | Baseline, Week 104
Time to First Occurrence of Any Component Event of the Composite Endpoint of Major Adverse Cardiovascular Events (MACE-3) | Baseline up to Study Completion (about 224 weeks)
  MACE-3 composite endpoint includes nonfatal myocardial infarction, nonfatal stroke, cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (556):
- United States (140):
  - MFA Clinical Research, Tuscaloosa, Alabama
  - The Institute for Liver Health II dba Arizona Clinical Trials - Chandler, Chandler, Arizona
  - Spectrum Research Institute, Gilbert, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health - Peoria, Peoria, Arizona
  - Epic Medical Research-Sun City, Sun City, Arizona
  - The Institute for Liver Health II dba Arizona Clinical Trials - Tucson, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Arkansas Gastroenterology - North Little Rock, North Little Rock, Arkansas
  - San Fernando Valley Health Institute, Canoga Park, California
  - Ark Clinical Research - Fountain Valley, Fountain Valley, California
  - Fresno Clinical Research Center, Fresno, California
  - UCSD - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - Orange County Research Center, Lake Forest, California
  - Om Research LLC, Lancaster, California
  - Ark Clinical Research, Long Beach, California
  - Los Angeles Institute for Metabolic Research, Los Angeles, California
  - United Medical Doctors - Murrieta, Murrieta, California
  - Knowledge Research Center, Orange, California
  - California Liver Research Center, Pasadena, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - K2 Medical Research WINTER GARDEN, Clermont, Florida
  - K2 Medical Research - Daytona Beach, Daytona Beach, Florida
  - Care Access - Delray Beach, Delray Beach, Florida
  - AMR Clinical, Doral, Florida
  - Southwest General Healthcare Center, Fort Myers, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Encore Medical Research, Hollywood, Florida
  - Nature Coast Clinical Research - Inverness, Inverness, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - Health Awareness, Jupiter, Florida
  - K2 MEDICAL Research THE VILLAGES, Lady Lake, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Tampa Bay Medical Research - Largo, Largo, Florida
  - Evolution Clinical Trials, Miami, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - GI PROS Research, Naples, Florida
  - Charter Research - Orlando, Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Metabolic Specialists - Riverview, Riverview, Florida
  - Care Access - St. Petersburg, St. Petersburg, Florida
  - Care Access - Tamarac, Tamarac, Florida
  - Covenant Metabolic Specialists, LLC, University Park, Florida
  - Southeast Clinical Research Center, Dalton, Georgia
  - Teak Research Consults, Lawrenceville, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Gastroenterology Health Partners, New Albany, Indiana
  - Deaconess Clinic- Gateway, Newburgh, Indiana
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - AMR Clinical, El Dorado, Kansas
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - AMR Clinical, Lexington, Kentucky
  - Delta Research Partners of Bastrop, LLC, Bastrop, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Care Access - New Iberia, New Iberia, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Delta Research Partners of West Monroe, West Monroe, Louisiana
  - Mercy Medical Center - Baltimore, Baltimore, Maryland
  - Capital Digestive Care - Chevy Chase, Chevy Chase, Maryland
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Clinton Township, Michigan
  - Great Lakes Research Institute, Southfield, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - MNGI Digestive Health, Minneapolis, Minnesota
  - GI Associates - GIA and Endoscopy Center - Flowood, Flowood, Mississippi
  - AMR Clinical, Kansas City, Missouri
  - Jubilee Clinical Research NV. LLC, Las Vegas, Nevada
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Advanced Research Institute - Reno, Reno, Nevada
  - Tandem Clinical Research - Freehold, Freehold, New Jersey
  - Atlantic Health System Morristown Medical Center, Morristown, New Jersey
  - Clinical Research of Philadelphia, Pennington, New Jersey
  - The Cognitive and Research Center of New Jersey - Ridgewood, Ridgewood, New Jersey
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Southwest Gastroenterology Associates, Albuquerque, New Mexico
  - Research Foundation of SUNY - University of Buffalo, Buffalo, New York
  - NYU Langone Health, New York, New York
  - IMA Clinical Research Manhattan, New York, New York
  - New York Gastroenterology Associates, New York, New York
  - Care Access - Yonkers, Yonkers, New York
  - Duke University - Main Hospital and Clinics, Durham, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Akron Gastro Research, Akron, Ohio
  - Dayton Gastroenterology - Beavercreek, Beavercreek, Ohio
  - CRIOH, Westlake, Ohio
  - US Digestive Health - Flourtown, Flourtown, Pennsylvania
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - US Digestive Health - Wyomissing, Wyomissing, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Columbia Digestive Health Research, Columbia, South Carolina
  - Galen Medical Group - Galen Hepatology, Chattanooga, Tennessee
  - Gastro One (Walnut Run Road), Cordova, Tennessee
  - American Research Corporation at Texas Liver Institute, Austin, Texas
  - IMA Clinical Research Austin, Austin, Texas
  - American Research Corporation, Austin, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - Bellaire Clinical Research, Bellaire, Texas
  - South Texas Research Institute - Brownsville, Brownsville, Texas
  - Headlands Horizons, LLC dba Headlands Research-Brownsville, Brownsville, Texas
  - Soma Clinical Trials, Denison, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - DHR Health Institute for Research and Development (Administrative Office & Laboratory), Edinburg, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Dallas Research Institute, Farmers Branch, Texas
  - Care United Research, LLC, Forney, Texas
  - GI Alliance - Fort Worth, Fort Worth, Texas
  - HRI- Medical Center, Houston, Texas
  - Care Access - Houston, Houston, Texas
  - Houston Research Institute, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - HRI Pasadena, Pasadena, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - GI Alliance - Southlake, Southlake, Texas
  - Houston Research Institute (HRI) - Sugar Land, Sugar Land, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Medrasa Clinical Research, Wylie, Texas
  - Care Access - Ogden, Ogden, Utah
  - Advanced Research Institute - Sandy, Sandy City, Utah
  - Eximia Research - Norfolk, Norfolk, Virginia
  - Richmond Veterans Affairs Medical Center (Richmond VA Medical Center), Richmond, Virginia
  - Gastroenterology Consultants of Southwest Virginia, Roanoke, Virginia
  - Washington Gastroenterology - Bellevue, Bellevue, Washington
  - UW Medicine Diabetes Institute, Seattle, Washington
  - Washington Gastroenterology - Tacoma, Tacoma, Washington
  - CAMC Health Education and Research Institute Inc, Charleston, West Virginia
- Argentina (17):
  - Hospital Italiano de Buenos Aires, ABB
  - CIPREC, Buenos Aires
  - DOM Centro de Reumatología, Buenos Aires
  - Glenny Corp. S.A., Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata
  - DIM Clínica Privada, Ramos Mejía
  - INECO Neurociencias Oroño, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Centro de Diagnóstico y Rehabilitación (CEDIR), Santa Fe
- Australia (15):
  - Nightingale Research, Adelaide
  - Flinders Medical Centre, Adelaide
  - Box Hill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Core Research Group, Brisbane
  - Mater Misericordiae Limited, Brisbane
  - Gallipoli Medical Research Ltd, Brisbane
  - Genesis Research Services, Broadmeadow
  - Austin Health, Heidelberg
  - Ipswich Hospital, Ipswich
  - Fiona Stanley Hospital, Murdoch
  - TrialsWest - Osborne Park, Osborne Park
  - The Royal Melbourne Hospital, Parkville
  - Gold Coast University Hospital, Southport
  - Westmead Hospital, Westmead
- Austria (5):
  - Medizinische Universität Graz, Graz
  - Uniklinikum Salzburg, Salzburg
  - Klinik Landstraße, Vienna
  - Medizinische Universität Wien, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (11):
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - AZ Oostende vzw, Ostend
  - AZ Delta vzw, Roeselare
  - VITAZ, Sint-Niklaas
- Brazil (27):
  - NewData Clinical Research - Aracaju, Aracaju
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - Hospital Universitário João de Barros Barreto, Belém
  - NUPEC - Cardio, Belo Horizonte
  - Faculdade de Medicina da UNESP, Botucatu
  - Centro de Pesquisa Clinica do Brasil, Brasília
  - Chronos Pesquisa Clínica, Brasília
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Cline Research Center, Curitiba
  - Hospital Universitario Walter Cantidio, Fortaleza
  - Universidade Federal de Goias, Goiânia
  - Hospital Brasilia, Lago Sul
  - CHN - Complexo Hospitalar de Niterói, Niterói
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital Moinhos de Vento, Porto Alegre
  - IMV Pesquisa Cardiologica - Porto Alegre - Rua Orfanotrofio, Porto Alegre
  - Instituto do Fígado e Tranplantes de Pernambuco, Recife
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Escola Bahiana de Medicina e Saúde Pública, Salvador
  - Inovace Pesquisa Clínica, Salvador
  - Centro Multidisciplinar de Estudos Clinicos, São Bernardo do Campo
  - CPHosp Medicina, Ensino e Pesquisa (CPQuali), São Paulo
  - Clínica Hepatogastro JK, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
  - CEDOES, Vitória
- Bulgaria (3):
  - University Hospital "St. Ivan Rilski", Gorna Oryahovitsa
  - Saint Marina Hospital, Pleven
  - UMHATEM 'N.I. Pirogov', Sofia
- Canada (14):
  - Heritage Medical Research Clinic, Calgary
  - Ecogene-21, Chicoutimi
  - Wells Research Group, Edmonton
  - University Of Alberta Hospital, Edmonton
  - University Hospital - London Health Sciences Centre, London
  - Private Practice - Dr. Stephane M. Gauthier, North Bay
  - Diex Recherche Quebec, Québec
  - Clinical Research of Ontario, Toronto
  - Toronto General Hospital, Toronto
  - St. Joseph's Health Centre, Toronto
  - Diex Recherche Inc. Division Trois-Rivieres, Trois-Rivières
  - Vancouver General Hospital, Vancouver
  - (G.I.R.I.) GI Research Institute Foundation, Vancouver
  - Health Sciences Centre Winnipeg, Winnipeg
- China (43):
  - Beijing Ditan Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing
  - Beijing Youan Hospital, Beijing
  - Hunan Provincial People's Hospital, Changsha
  - Xiangya Hospital Central South University, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - 2nd Affiliated Hospital Chongqing Medical University, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - Fujian Medical University Mengchao Hepatobiliary Hospital (Fuzhou Infectious Disease Hospital), Fuzhou
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - Guangzhou 8th People's Hospital, Guangzhou
  - Southern Medical University Nanfang Hospital, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - Jinhua Central Hospital, Jinhua
  - Liaocheng People's Hospital, Liaocheng
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - The Affiliated Hospital of Southwest Medical University, Luzhou
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The First affiliated hospital of Nanchang University (Xianghu campus), Nanchang
  - Jiangsu Province Hospital, Nanjing
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - Ningbo 2nd Hospital, Ningbo
  - The first affiliated hospital of Ningbo university, Ningbo
  - Ningbo Medical Center, Ningbo
  - Pingxiang People's Hospital, Pingxiang
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital,Fudan University, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin People' s Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
  - Zhoukou Central Hospital, Zhoukou
- Czechia (3):
  - Krajská nemocnice Liberec, Liberec
  - Fakultni nemocnice Ostrava, Ostrava
  - Mestska nemocnice Ostrava, Ostrava
- France (16):
  - CHU d'Amiens-Picardie - Hôpital Sud, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - CHU Besançon, Besançon
  - Hôpital Beaujon, Clichy
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - CHD Vendee, La Roche-sur-Yon
  - Hopital Claude Huriez - CHU de Lille, Lille
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Pitie Salpetriere University Hospital, Paris
  - Hôpital Saint Antoine, Paris
  - CHU Bordeaux Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes
  - CHU Rangueil, Toulouse
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux
- Germany (13):
  - Herz - und Diabeteszentrum Nordrhein - Westfalen, Bad Oeynhausen, Bad Oeynhausen
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden
  - Deutsches Diabetes-Zentrum (DDZ), Düsseldorf
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Eugastro GmbH, Leipzig
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz
  - Ruppiner Kliniken, Neuruppin
- Hungary (3):
  - Óbudai Egészségügyi Centrum, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház, Nyíregyháza
- India (20):
  - Avron Hospitals, Ahmedabad
  - All India Institute of Medical Sciences, Bhubaneswar
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Amrita Institute of Medical Sciences and Research Center, Ernākulam
  - Asian Institute of Gastroenterology, Hyderabad
  - SR Kalla Memorial Gastro & General Hospital, Jaipur
  - Lisie Hospital, Kochi
  - John C. Martin Centre for Liver Research & Innovations (JCMLRI), Kolkata
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow
  - Dayanand Medical College and Hospital, Ludhiana
  - Fortis Hospital - Mohali, Mohali
  - Topiwala National Medical College & B. Y. L. Nair Charitable Hospital, Mumbai
  - Mysore Medical College, Mysore
  - Midas Multispeciality Hospital Pvt.Ltd., Nagpur
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - All India Institute of Medical Sciences - Rishikesh, Rishikesh
  - Surat Institute of Digestive Sciences Hospitals, Surat
  - Acharya Vinoba Bhave Rural Hospital, Wardha
- Israel (11):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Carmel Hospital, Haifa
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Maccabi Health Services - Petah Tikva, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
  - Assuta Medical Center, Tel Aviv
- Italy (11):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Federico II, Naples
  - Azienda Ospedale - Università Padova, Padua
  - A.O.U. Policlinico Paolo Giaccone, Palermo
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
- Japan (63):
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki
  - Asahikawa Medical University Hospital, Asahikawa
  - Institute of Science Tokyo Hospital, Bunkyō
  - Juntendo University Hospital, Bunkyō City
  - The University of Tokyo Hospital, Bunkyō City
  - Tokyo Metropolitan Komagome Hospital, Bunkyō City
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Hamanomachi Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Gifu Municipal Hospital, Gifu
  - University of the Ryukyus Hospital, Ginowan
  - Hamamatsu University Hospital, Hamamatsu
  - Hiroshima University Hospital, Hiroshima
  - National Kohnodai Medical Center, Ichikawa
  - Nihon University Itabashi Hospital, Itabashiku
  - Shimane University Hospital, Izumo
  - Juntendo University Shizuoka Hospital, Izunokuni
  - Kagoshima University Hospital, Kagoshima
  - Nara Medical University Hospital, Kashihara
  - St. Marianna University Hospital, Kawasaki
  - Kagawa University Hospital, Kita-ku
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kumamoto University Hospital, Kumamoto
  - Kumamoto Shinto General Hospital, Kumamoto
  - Kurume University Hospital, Kurume
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Saiseikai Maebashi Hospital, Maebashi
  - Toranomon Hospital, Minatoku
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Japanese Red Cross Musashino Hospital, Musashino-shi
  - Nagasaki University Hospital, Nagasaki
  - Meitetsu Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - International University of Health and Welfare Narita Hospital, Narita
  - Hyogo Medical University Hospital, Nishinomiya
  - Okayama University Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Keisatsu Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Abe Clinic, Ōita
  - Oita Cardiovascular Hospital, Ōita
  - National Hospital Organization Nagasaki Medical Center, Ōmura
  - Saga University Hospital, Saga
  - Osaka Rosai Hospital, Sakai
  - Bell Land General Hospital, Sakai
  - Hokkaido University Hospital, Sapporo
  - Jichi Medical University Hospital, Shimotsuke
  - National Center for Global Health and Medicine, Shinjyuku-ku
  - Iwate Medical University Hospital, Shiwa-gun Yahaba-cho
  - Osaka Saiseikai Suita hospital, Suita
  - The University of Osaka Hospital, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - National Hospital Organization Takasaki General Medical Center, Takasaki
  - Tokyo Women's Medical University, Tokyo
  - Nagano Municipal Hospital, Tomitake
  - Sekino Hospital, Toshimaku
  - Ehime University Hospital, Tōon
  - Mie University Hospital, Tsu
  - National Hospital Organization Ureshino Medical Center, Ureshino
  - Yamagata University Hospital, Yamagata
  - Yokohama City University Hospital, Yokohama
- Malaysia (2):
  - Hospital Universiti Sains Malaysia, Kubang Kerian
  - University Malaya Medical Centre, Lembah Pantai
- Mexico (17):
  - Medical Center Metas, Chihuahua City
  - Centro de Investigación y Gastroenterología, Cuauhtémoc
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca
  - Centro de Investigación Clínica y Medicina Traslacional (CIMeT), Guadalajara
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara
  - Unidad de Investigación Clínica y Atención Médica HEPA S.C., Guadalajara
  - Centro Médico Lic. Arturo Montiel Rojas ISSEMYM, Metepec
  - Grupo Medico Camino Sc, Mexico City
  - Centro de Investigación y Gastroenterología - S.C., Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - CEINV Salud, Monterrey
  - Clinica de Enfermedades Cronicas y Procedimientos Especiales, SC, Morelia
  - Oncare Vasconcelos, San Pedro Garza García
  - Avant Sante Research Center, San Pedro Garza García
  - Fundación Santos y de la Garza Evía I.B.P, San Pedro Garza García
  - Hospital General de Occidente, Zapopan
- Netherlands (5):
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- New Zealand (3):
  - New Zealand Clinical Research (Auckland), Auckland
  - Aotearoa Clinical Trials, Auckland
  - Aotearoa Clinical Trials - Whangarei, Whangarei
- Norway (2):
  - Oslo Universitetssykehus Ullevål, Oslo
  - Universitetssykehuset Nord-Norge HF, Tromsø
- Poland (15):
  - KRESMED Sp. z o.o., Bialystok
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk
  - Centrum Medyczne Pratia Katowice, Katowice
  - Gyncentrum sp. z o.o. NZOZ Holsamed - oddział Libero, Katowice
  - Santa Familia PTG Lodz, Lodz
  - ID Clinic, Mysłowice
  - Uniwersyteckie Centrum Stomatologii i Medycyny Specjalistycznej, Poznan
  - Private Practice - Dr. Lukasz Krupa, Rzeszów
  - NZOZ GynCentrum - Oddział Warszawa, Warsaw
  - Przychodnie Care Access, Warsaw
  - Szpital Czerniakowski, Warsaw
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - Państwowy Instytut Medyczny MSWiA, Warsaw
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw
  - ETG Zamość, Zamość
- Portugal (2):
  - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
- Puerto Rico (2):
  - Isis Clinical Research Center, Guaynabo
  - Klinical Investigations Group, San Juan
- Romania (5):
  - Delta Health Care, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Regional de Gastroenterologie și Hepatologie Prof. Dr. Octavian Fodor, Cluj-Napoca
  - Constanta County Emergency Clinical Hospital Sf.Ap.Andrei, Constanța
  - Spital Judetean de Urgenta, Satu Mare
- South Korea (19):
  - Korea University Ansan Hospital, Ansan-si
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si
  - Pusan National University Yangsan Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Chung-Ang University Hospital, Dongjak-gu
  - Boramae Medical Center, Dongjak-gu
  - Hanyang University Guri Hospital, Guri-si
  - Yeungnam Univeristy Medical Center, Gyeongsan-si
  - Inha University Hospital, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Kyungpook National University Hospital, Junggu
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Spain (13):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol
  - Hospital Infanta Elena, Huelva
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari Son Espases, Palma
  - CHOP - Hospital Universitario Montecelo, Pontevedra
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (2):
  - Karolinska Universitetssjukhuset Huddinge, Huddinge
  - Universitetssjukhuset i Linköping, Linköping
- Switzerland (3):
  - University Hospital Basel, Basel
  - Luzern Kantonsspital, Lucerne
  - Kantonsspital Olten, Olten
- Taiwan (15):
  - Chiayi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - Taipei Tzu Chi General Hospital, New Taipei City
  - Fu Jen Catholic University Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (8):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Çukurova Üniversitesi Tıp Fakültesi Adana Hastanesi, Adana
  - Hacettepe Universitesi, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Bursa Şehir Hastanesi, Bursa
  - T.C. Sağlik Bakanliği- Marmara Üniversitesi İstanbul Pendik Eğitim Ve Araştirma Hastanesi, Pendik
  - Recep Tayyip Erdogan University Training and Research Hospital, Rize
  - Karadeniz Teknik Universitesi Tip Fakultesi, Trabzon
- Ukraine (11):
  - Clinical Diagnostic Center, Ivano-Frankivsk
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kiev
  - Edelweiss Medics, Kyiv
  - Medical Center Ok!Clinic+, Kyiv
  - Medbud Clinic, Kyiv
  - Center of Family Medicine Plus, Kyiv
  - Progastro Clinic, Lviv
  - Medical Center Salutem, Vinnytsia
  - Limited liability company "Medical center Health Clinic", Vinnytsia
  - Municipal Nonprofit Enterprise "Vinnytsia Regional Clinical Hospital n.a. M. I. Pyrohov of Vinnytsia Regio -T, Vinnytsia
  - CRZ Vidnovlennya, Zhytomyr
- United Kingdom (17):
  - Aberdeen Royal Infirmary, Aberdeen
  - 4 Medical Solutions, Ltd - Manchester, Clifton
  - Panthera Biopartners - North London, Enfield
  - Panthera Biopartners - Glasgow, Glasgow
  - Ipswich Hospital, Ipswich
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Royal London Hospital, London
  - 4 Medical Solutions, Ltd - London, London
  - Royal Free Hospital, London
  - King's College Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - The John Radcliffe Hospital, Oxford
  - Panthera Biopartners - Preston, Preston
  - Panthera Biopartners - Manchester, Rochdale
  - Panthera Biopartners - Sheffield, Sheffield
  - Musgrove Park Hospital, Taunton
  - Panthera Clinic - York, York

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Master Protocol of Multiple Agents in Adults With Metabolic Dysfunction-Associated Steatotic Liver Disease (SYNERGY-Outcomes) — https://trials.lilly.com/en-US/trial/651596